CLINICAL TRIAL: NCT01666704
Title: A Double-Blind, Placebo-Controlled, Randomized Study to Evaluate the Effects of BMS-823778 on Atherosclerotic Plaque Inflammation as Measured by Fluorodeoxyglucose (FDG)- Positron Emission Tomography (PET) in Patients With Atherosclerotic Cardiovascular Disease
Brief Title: Proof of Concept Study of BMS-823778 to Assess the Effects on Atherosclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB121-010
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — BMS-823778

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A: BMS-823778 (2mg) (Experimental)
  Interventions: Drug: BMS-823778
- Treatment B: BMS-823778 (15mg) (Experimental)
  Interventions: Drug: BMS-823778
- Treatment C: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching with BMS-823778

INTERVENTIONS:
Drug: BMS-823778 — Capsules, Oral, 2mg, Once daily, 1 year
  Arms: Treatment A: BMS-823778 (2mg)
Drug: BMS-823778 — Capsules, Oral, 15mg, Once daily, 1 year
  Arms: Treatment B: BMS-823778 (15mg)
Drug: Placebo matching with BMS-823778 — Capsules, Oral, 0mg, Once daily, 1 year
  Arms: Treatment C: Placebo

SUMMARY:
The purpose of the study is to assess the effect of BMS-823778 on reducing atherosclerotic plaque inflammation

ELIGIBILITY:
Inclusion Criteria:

* Documented atherosclerotic cardiovascular disease or at high risk of cardiovascular event
* On stable statin dose
* Clinically stable at time of screening and randomization

Exclusion Criteria:

* Women of child bearing potential
* Medical conditions that would impact the absorption of the study drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2015-10 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
The effect of BMS-823778 versus placebo on carotids and/or ascending aortic will be measured by fluorodeoxyglucose (FDG) uptake in the index vessel as by positron emission tomography (PET) imaging | Day 168

SECONDARY OUTCOMES:
Structural changes in the arterial wall (absolute, percent change, and both, from baseline in four indices) | Day 364
  Structural changes in the arterial wall (absolute, percent change, and both, from baseline in four indices): total vessel area, wall area, wall thickness, and wall area/total vessel area ratio (normalized wall index), based on the average of the right and left carotids, measured by Magnetic Resonance Imaging (MRI)
Safety will be measured by adverse event, vital signs, electrocardiogram, physical examinations, clinical laboratory tests and Ferriman- Gallwey scores | Approximately up to 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx